CLINICAL TRIAL: NCT01807715
Title: Understanding Women's Contraceptive Expectations at the Time of a First Trimester Surgical Abortion
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 352286
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Contraception; Abortion
Keywords: first trimester; surgical abortion; contraception
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Women seeking first trimester surgical abortion
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — Survey before procedure to obtain demographic information and contraceptive information

SUMMARY:
The investigators will conduct a voluntary anonymous survey at four separate Sacramento area family planning clinics. The investigators will ask the staff at each facility to offer a survey to all women 18 and older presenting to the clinic to have a first trimester (<12 weeks gestation) surgical abortion. Gestational age will be based on what the woman believes is her gestational age at presentation, before any evaluation in the clinic. Women who cannot understand or read the survey will be excluded. The investigators hope to implement the survey at these clinics for 3-4 months reaching a minimum of 200 women (based on a target population of 600 women receiving surgical first trimester abortions at these two clinics over a 3-4 month period with a 95% confidence interval).

DETAILED DESCRIPTION:
We will conduct a voluntary anonymous survey at four separate Sacramento area family planning clinics. We will introduce the research project to clinic staff, recruiting their support and participation, as they will be the main implementers. The survey will be offered to women in the waiting room before any pre-procedure counseling. We will include all women presenting to the clinic who are 18 years and older and planning to have a first trimester (<12 weeks gestation) surgical abortion. Gestational age will be based on what the woman believes is her gestational age at presentation, before any evaluation in the clinic. Women who cannot understand or read the survey will be excluded. We hope to implement the survey at these two clinics for 3-4 months reaching a minimum of 200 women so as to obtain an adequate power for our study. The brief survey will include a cover letter explaining the study and stressing the anonymity and confidentiality. The surveys will include an envelope in which to place completed surveys; the envelope can be sealed by the participant and dropped in a collection bin. This process will allow the data to be collected anonymously. The survey data will then be synthesized first by descriptive analysis, followed by chi-square and multiple regression analyses. A statistician in the University of California Davis Department of Obstetrics and Gynecology will help when necessary.

ELIGIBILITY:
Inclusion Criteria:

* seeking first trimester surgical abortion

Exclusion Criteria:

* Women who cannot understand or read the survey

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women seeking first trimester surgical abortion
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
patient preference | one day
  patient preference for whether she wants to discuss contraception during her visit for an abortion

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell D Creinin, MD, Study Director — UC Davis; Melissa Matulich, Principal Investigator — UC Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Matulich M, Cansino C, Culwell KR, Creinin MD. Understanding women's desires for contraceptive counseling at the time of first-trimester surgical abortion. Contraception. 2014 Jan;89(1):36-41. doi: 10.1016/j.contraception.2013.09.013. Epub 2013 Sep 30. PMID 24161475